CLINICAL TRIAL: NCT00814281
Title: Airborne Ultrafine and Fine Particulate Matter: A Cause for Endothelial Dysfunction in Man?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marywood University (Other)
Responsible Party: Kenneth W. Rundell Ph.D., Marywood University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MU2007-005
Record Dates: First submitted 2008-12-22; First posted 2008-12-24 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Airway Inflammation
Keywords: particulate air pollution; leukotriene; asthma; montelukast; vascular endothelial dysfunction; nitric oxide(NO)endothelin (ET) system
MeSH Terms: conditions — Asthma | interventions — Sugars; montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Subject will exercise in high levels of ultrafine and fine particulate air pollution 1 hour after ingesting a placebo.
  Interventions: Other: placebo
- 2 (Placebo Comparator): Subject will exercise in low levels of ultrafine and fine particulate air pollution 1 hour after ingesting a placebo.
  Interventions: Other: placebo
- 3 (Experimental): Subject will exercise in high levels of ultrafine and fine particulate air pollution 1 hour after ingesting Montelukast 10 mg orally.
  Interventions: Drug: Montelukast
- 4 (Experimental): Subject will exercise in low levels of ultrafine and fine particulate air pollution 1 hour after ingesting Montelukast 10 mg orally.
  Interventions: Drug: Montelukast

INTERVENTIONS:
Other: placebo — Placebo
  Other Names: Sugar Pill
  Arms: 1; 2
Drug: Montelukast — 10 mg ingested orally 1 hour prior to exercise testing
  Other Names: Singulair
  Arms: 3; 4

SUMMARY:
The purpose of this study is to examine biological pathways of altered blood vessel function resulting from breathing airborne particulate. Blood artery function in healthy men will be measured after particulate exposure either on placebo or on an asthma medication that stops production of an inflammatory biological agent. Lung and blood profiles will be obtained before and after exposure to exhaust fumes. We believe that the inflammatory agent produced by the lungs from breathing these particles causes abnormal artery function.

DETAILED DESCRIPTION:
Hourly ice resurfacing by gas and propane fueled machines creates high levels of ultrafine and fine particulate matter (PM1) in indoor ice rinks. PM1 exposure may disrupt the normal nitric oxide (NO)/endothelin (ET)-1 vasodilation system and promote atherosclerosis, and/or increase the risk of an acute cardiac event. Our specific aims are 1) to determine whether impaired endothelial-mediated vasodilation and forearm muscle tissue reoxygenation rate and blood volume change (to reactive hyperemia following artery occlusion) is associated with combustion-derived PM1 exposure, and 2) To characterize a PM1 induced mechanism of endothelial dysfunction which occurs via a leukotriene (LT)-associated, airway generated tumor necrosis factor-alpha (TNF-a) mediated pathway. Healthy low PM1 exposed males will be evaluated for endothelial dysfunction before and after artery occlusion using high resolution ultrasound and near-infrared spectroscopy (NIRS), before and after moderate exercise in blinded high and low [PM1]. Endothelial dysfunction among chronically PM¬1 exposed ice rink athletes will be determined to evaluate the feasibility of using this population as a model in future studies. TNF-a, IL-8, LTB4, LTC4, LTD4, LTE4, ET-1, NO, and differential cell counts will be measured in sputum and serum. [PM1] will be monitored and exposure levels will be typical of indoor ice rinks. LT involvement will be assessed in vivo by double-blind pharmacological manipulation during PM1 exposure during light exercise. Results will demonstrate whether endothelial-mediated vasodilation and muscle hemodynamics are influenced by PM1 exposure, and will elucidate an LT initiated TNF-a mediated pathway in ET-1 upregulation. Our results should provide information for understanding the effects of PM1 exposure on the atherosclerotic process and cardiovascular risk, and give insight to novel treatment and diagnostic modalities.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* between 18 and 30 years of age
* participant in endurance sport

Exclusion Criteria:

* history of blood clotting
* history of coagulation problems
* History of spontaneous pneumothorax

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Exposure to airborne ultrafine and fine particulate matter causes vascular dysfunction. | February 2009

SECONDARY OUTCOMES:
Montelukast protects against pollution induced vascular dysfunction. | February 2009

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth W Rundell, PhD, Principal Investigator — Marywood University
Locations (1):
- Marywood University, Scranton, Pennsylvania, United States